CLINICAL TRIAL: NCT02610218
Title: Liquid Biopsy in Monitoring the Therapeutic Efficacy of Targeted Therapy in Advanced/Metastatic Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology, Peking University
Other Study IDs: LiquidBiopsy
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Gastric Cancer
Keywords: Cell free DNA; Circulating tumor cell; Therapeutic efficacy
MeSH Terms: conditions — Stomach Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples of 12.5 mL were collected from the patients for cfDNA and CTCs analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- histo-HER2+ gastric cancer patients: Histologically HER2 positive gastric cancer patients treated with HER2 targeted therapy. Interventions: peripheral blood samples of 12.5 mL for CTC and cfDNA analysis will be collected before targeted therapy, at the time that they achieve the optimal response and when they suffer progressive disease.
  Interventions: Other: CTC and cfDNA analysis
- histo-HER2- gastric cancer patients: Histologically HER2 negative gastric cancer patients treated with chemotherapy. Interventions: peripheral blood samples of 12.5 mL for CTC and cfDNA analysis will be collected before targeted therapy, at the time that they achieve the optimal response and when they suffer progressive disease.
  Interventions: Other: CTC and cfDNA analysis

INTERVENTIONS:
Other: CTC and cfDNA analysis — The enumeration of CTCs as well as the detection of HER2 expression will be achieved via the integrated subtraction enrichment (SET) and immunostaining-fluorescence in situ hybridization (iFISH) platform. Further, for the geneomic analysis, the enriched single CTC will be isolated for single-cell targeted sequencing. While for cfDNA analysis, extracted DNA from plasma will be directly subjected to targeted sequencing. Tumor response evaluation will be performed after two cycles of chemotherapy by CT/MRI based on RECIST. Clinical data, including tumor stage, metastastic organ, chemotherapy regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
To evaluate the clinical significance of cell free DNA (cfDNA) and circulating tumor cells (CTCs) in real-time monitoring the therapeutic response during HER2-targeted therapy in histologically confirmed HER2 positive advanced/metastatic gastric cancer.

DETAILED DESCRIPTION:
The study is a single-center, prospective study undertaken in anticipated 124 patients with both histologically HER2 positive and negative advanced/metastatic gastric cancer. Peripheral blood samples of 12.5 mL were collected from the patients for cfDNA and CTCs analysis. The blood samples will be respectively drawn before therapy, at the time that the patients achieve the optimal response and when they suffer progressive disease. The enumeration of CTCs as well as the detection of HER2 expression will be achieved via the integrated subtraction enrichment (SET) and immunostaining-fluorescence in situ hybridization (iFISH) platform. Further, for the geneomic analysis, the enriched single CTC will be isolated for single-cell targeted sequencing. While for cfDNA analysis, extracted DNA from plasma will be directly subjected to targeted sequencing. The correlation of the HER2 status on CTCs and the HER2 amplification in cfDNA to the therapeutic response will be evaluated. Moreover, gene variations associated with resistance in HER2-targeted therapy will be also studied based on the genomic data from sequencing of CTC and cfDNA.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed HER2 positive gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥60
* Life expectancy of ≥2 month
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <ULN, and CCr < 60ml/min
* Bilirubin level < 1.5 ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Brain metastasis (known or suspected)
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry. Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
* Allergic constitution or allergic history to protium biologic product or any investigating agents.
* Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Pre-existing neuropathy>grade 1
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anticipated 124 patients with histologically confirmed HER2 positive advanced/metastatic gastric cancer
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of HER2 status on CTCs and cfDNA with clinical outcomes | through study completion, an average of 1 year
  To evaluate the correlation of CTCs and their HER2 expression status to the clinical outcomes

SECONDARY OUTCOMES:
Gene variations associated with resistance in HER2-targeted therapy | up to 6 months
  To study the gene variations associated with resistance in HER2-targeted therapy based on the genomic data from sequencing of CTC and cfDNA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of GI Oncology, Peking University Cancer Hospital, Beijing, Beijing Municipality, China